CLINICAL TRIAL: NCT06395662
Title: Improving the Stratification of Risks of Conversion of Radiologically Isolated Syndromes (RIS) by Identifying Biomarkers in Serum and Cerebrospinal Fluid. The ProBioRIS Study
Brief Title: Stratification of Risks of Conversion of Radiologically Isolated Syndromes (RIS) by Identifying Biomarkers in Serum and Cerebrospinal Fluid.
Acronym: ProBioRIS
Status: Active, not recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Collaborators: International Center of Research in Infectiology, Lyon University (Unknown); Universite Cote d'Azur (Other); The University of Texas at Dallas (Other)
Responsible Party: Sponsor
Other Study IDs: ProBioRIS
Record Dates: First submitted 2024-04-29; First posted 2024-05-02 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Radiologically Isolated Syndrome; Multiple Sclerosis
Keywords: Radiologically Isolated Syndrome; Multiple Sclerosis; Biomarkers
MeSH Terms: conditions — Multiple Sclerosis | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biological samples and magnetic resonance imaging data from four large cohorts of patients with multiple sclerosis in the United States, Europe and France will be used for this study. Indeed, this proposal is based on existing clinical and magnetic resonance imaging data and stored serum and cerebrospinal fluid samples from ARISE (clinicaltrials. gov NCT02739542) and TERIS (NCT03122652), which are randomized, double-blind, placebo-controlled trials in multiple sclerosis, as well as two prospective, real-world cohorts of multiple sclerosis patients from the French multiple sclerosis registry (OFSEP) and the French multiple sclerosis society (SFSEP).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- ARISE cohort: n=87, clinicaltrials.gov NCT02739542
  Interventions: Other: Observational
- TERIS cohort: n=90, clinicaltrials.gov NCT03122652
  Interventions: Other: Observational
- OFSEP cohort: OFSEP, n=75
  Interventions: Other: Observational
- SFSEP cohort: SFSEP, n=75
  Interventions: Other: Observational
- Subset of serum and cerebrospinal biomarkers: As a validation group, the best subset of serum and cerebrospinal biomarkers from Objective 2a will be tested in a separate group of RIS patients. Their association with the same outcomes (clinical relapse and magnetic resonance imaging measurements of disease severity/activity) will be measured using the same regression techniques as in Objective 2a. This subset will consist of the remaining third of RIS patients from the SFSEP, OFSEP, and ARISE cohorts with serum and cerebrospinal fluid available (n=60)
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Search for biomarkers

SUMMARY:
Radiologically isolated syndrome (RIS) often precedes Multiple Sclerosis (MS) but some patients have no symptoms. This study aims to use biological samples and magnetic resonance imaging (MRI) data from four large cohorts of patients with MS in the United States, Europe and France, to stratify the chances of RIS developing into MS. Identifying early biomarkers to predict greater disease severity would have a significant impact, not only on RIS but also on the entire clinical spectrum of multiple sclerosis.

DETAILED DESCRIPTION:
Radiologically Isolated Syndrome (RIS) is defined as the presence of asymptomatic, idiopathic demyelinating-appearing white matter lesions in the central nervous system. RIS often precedes clinical multiple sclerosis. Data from the international RIS Consortium indicate that 34% of RIS patients will have their first multiple sclerosis symptom within 5 years, and 51% within 10 years, making RIS the earliest identifiable phase of MS. While most RIS patients will evolve to relapsing MS, ~10% directly evolve towards progressive multiple sclerosis. RIS is an informative cohort for studying the earliest pathophysiologic changes, but remains a significant challenge for MS clinicians, as not all RIS patients will develop clinical symptoms. There is a need to distinguish RIS patients at high risk of clinical MS from those who will remain asymptomatic. Stratification would be invaluable to inform treatment/monitoring recommendations and counsel patients.

In the RIS Consortium cohort, age at diagnosis, positive CSF oligoclonal bands (OCBs) or elevated IgG index, infratentorial or spinal cord lesions, and gadolinium-enhancing (Gd+) lesions during follow-up independently predicted a first clinical event at 10 years. Additional serum and CSF biomarkers may further refine the risk stratification for clinical MS and may predict more severe tissue injury measured by MRI.

Serum and cerebrospinal fluid biomarkers can refine risk stratification of the progression from risk to clinical multiple sclerosis and predict more severe tissue damage as measured by magnetic resonance imaging. Identifying early biomarkers to predict greater disease severity would have a significant impact, not only on RIS, but also on the entire clinical spectrum of multiple sclerosis. However, RIS remains a rare disease and large cohorts are needed to validate potential prognostic biomarkers.

The international RIS Consortium has had a unique opportunity to apply for a research grant from the National Multiple Sclerosis Society to combine biomarker expertise, advanced magnetic resonance imaging analysis, and collaborative networks and cohorts to refine the prognosis of multiple sclerosis. Here, the proposal is to use biological samples and magnetic resonance imaging data from four large cohorts of patients with multiple sclerosis in the United States, Europe and France. In fact, this proposal is based on existing clinical and magnetic resonance imaging data and stored serum and cerebrospinal fluid samples from the ARISE (clinicaltrials. gov NCT02739542) and TERIS (NCT03122652) trials, which are randomized, double-blind, placebo-controlled trials on multiple sclerosis, as well as two prospective, real-world cohorts of multiple sclerosis patients from the French multiple sclerosis observatory (OFSEP = Observatoire Français de la Sclérose en Plaques) and the French multiple sclerosis society (SFSEP = Société Francophone de la Sclérose En Plaques).

The French observatory for multiple sclerosis, coordinated by Professor Sandra Vukusic in Lyon, brings together neurologists from all over France and 61 centers that use the European Database for Multiple Sclerosis, including 31 French hospitals and expert centers, and more than 45,000 people with multiple sclerosis or related diseases (half the population with multiple sclerosis in France). This includes a priority effort involving at least 85 RIS patients validated by the central supervision of the RIS consortium (Prof. Christine Lebrun-Frenay, Nice), with longitudinal follow-up and systematic association of clinical data with biological samples and neuro-imaging.

Standardized biological samples obtained from RIS patients and banked in certified biological resource centers guarantee the high quality of biological samples associated with clinical and medical imaging data collected prospectively in the EDMUS database. This biocollection offers a unique opportunity to identify and validate potential biomarkers of disease activity and clinical conversion in RIS patients, notably in association with those of randomized clinical trials and the SFSEP, which relies on the same French network of experts in multiple sclerosis (CRC-SEP = Centres de Ressources et de Compétences sur la Sclérose en Plaques) and biological research centers.

The hypothesis is that increases in the serum Neurofilament Light (sNfl) chain and serum Glial Fibrillary Astrocytic Protein (sGFAP) will be associated with higher numbers of new gadolinium-enhancing (Gd+) lesions, higher T2 lesion volume, higher rates of clinical relapse, and faster thalamic volume decline over 96 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients from the OFSEP, SFSEP, RISE and TERIS cohorts with centralized validated radiologoically isolated syndrome and a standardized magnetic resonance imaging from the OFSEP or Randomized Clinical Trials database.
* at least one cerebro-spinal fluid and/or serum sample at baseline available at a local or centralized biological resource center.
* if present, serum sample collected at the time of clinical conversion.

Exclusion Criteria:

* patients with no biocollection, or with non-standardized magnetic resonance imaging acquisitions

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All patients registered in the ARISE, TERIS, OFSEP and SFSEP cohorts.
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Aim 1a : Association between Serum Neurofilament Light chain (sNfL) and RIS in all groups of patients | Week 0
  Quantitative in g/mL, SIMOA (TM) in all cohorts: ARISE, TERIS, OFSEP and SFSEP. n=327
Aim 1a : Association between Serum Neurofilament Light chain (sNfL) and RIS in all groups of patients | Week 96
  Quantitative, in g/mL, SIMOA (TM) in all cohorts: ARISE, TERIS, OFSEP and SFSEP. n=327
Aim 1a : Association between Serum Glial Fibrillary Astrocytic Protein (sGFAP) and RIS in all groups of patients | Week 0
  Quantitative, in g/mL, SIMOA (TM) in all cohorts: ARISE, TERIS, OFSEP and SFSEP. n=327
Aim 1a : Association between Serum Glial Fibrillary Astrocytic Protein (sGFAP) and RIS in all groups of patients | Week 96
  Quantitative, in g/mL, SIMOA (TM) in all cohorts: ARISE, TERIS, OFSEP and SFSEP. n=327
Aim 1b: Association between Serum Neurofilament Light chain (sNfL) and RIS in placebo-treated patients | Week 0
  Serum Neurofilament Light chain (sNfL) will be measured in placebo-treated patients from the ARISE and TERIS cohorts (n= 88)
Aim 1b: Association between Serum Neurofilament Light chain (sNfL) and RIS in placebo-treated patients | Week 96
  Serum Neurofilament Light chain (sNfL) will be measured in placebo-treated patients from the ARISE and TERIS cohorts (n= 88)
Aim 1b : Association between Serum Glial Fibrillary Astrocytic Protein (sGFAP)and RIS in placebo-treated patients | Week 0
  Serum Glial Fibrillary Astrocytic Protein (sGFAP) will be measured in placebo-treated patients from the ARISE and TERIS cohorts (n= 88)
Aim 1b: Association between Serum Glial Fibrillary Astrocytic Protein (sGFAP)and RIS in placebo-treated patients | Week 96
  Serum Glial Fibrillary Astrocytic Protein (sGFAP)will be measured in placebo-treated patients from the ARISE and TERIS cohorts (n= 88)

SECONDARY OUTCOMES:
Aim 2a: Kappa free light chain (KFLC) index in RIS patients in the SFSEP, OFSEP and ARISE cohorts, n=121 | Week 0
  CSF NfL, CHI3L1, and OCBs have been tested as predictors of clinical evolution in RIS, but a comprehensive examination of a large number of candidate serum and CSF biomarkers has not been undertaken. The kappa free light chain (KFLC) index will be measured in two-thirds of the total cerebral spinal fluid samples available (n= 121) by cytokine multiplex assay (ProcartaPlexTM and Simoa TM). Regression techniques (chosen according to the outcome variable) will measure the univariate association between each CSF and serum biomarker and the number of Gd+ lesions, T2LV, and thalamic volume at study entry and new T2/Gd+ lesions, clinical relapse, and thalamic volume decline over time. Machine learning (LASSO; SAS HPGENSELECT) will select the final set of biomarkers most strongly associated with clinical and MRI measures.
Aim 2a: Kappa free light chain (KFLC) index in RIS patients in the SFSEP, OFSEP and ARISE cohorts, n=121 | Week 96
  CSF NfL, CHI3L1, and OCBs have been tested as predictors of clinical evolution in RIS, but a comprehensive examination of a large number of candidate serum and CSF biomarkers has not been undertaken. The kappa free light chain (KFLC) index will be measured in two-thirds of the total cerebral spinal fluid samples available (n= 121) by Binding Site Optilite analyzer. Regression techniques (chosen according to the outcome variable) will measure the univariate association between each CSF and serum biomarker and the number of Gd+ lesions, T2LV, and thalamic volume at study entry and new T2/Gd+ lesions, clinical relapse, and thalamic volume decline over time. Machine learning (LASSO; SAS HPGENSELECT) will select the final set of biomarkers most strongly associated with clinical and MRI measures.
Aim 2a: Cerebrospinal fluid neurofilament light chain as a potential biomarker of RIS. | Week 0
  The neurofilament light chain will be measured in two-thirds of the total cerebral spinal fluid samples available (n= 121) from patients in the SFSEP, OFSEP and ARISE cohorts by cytokine multiplex assay (Simoa TM).
Aim 2a: Cerebrospinal fluid neurofilament light chain as a potential biomarker of RIS. | Week 96
  The neurofilament light chain will be measured in two-thirds of the total cerebral spinal fluid samples available (n= 121) from patients in the SFSEP, OFSEP and ARISE cohorts by cytokine multiplex assay (Simoa TM).
Aim 2a: Chitinase-3-like protein 1 as a potential biomarker of RIS. | Week 0
  Chitinase-3-like protein 1will be measured in two-thirds of the total cerebral spinal fluid samples available (n= 121) from patients in the SFSEP, OFSEP and ARISE cohorts by cytokine multiplex assay (ProcartaPlexTM).
Aim 2a: Chitinase-3-like protein 1 as a potential biomarker of RIS. | Week 96
  Chitinase-3-like protein 1will be measured in two-thirds of the total cerebral spinal fluid samples available (n= 121) from patients in the SFSEP, OFSEP and ARISE cohorts by cytokine multiplex assay (ProcartaPlexTM).
Aim 2a: Oligoclonal bands as a potential biomarker of RIS. | Week 0
  Oligoclonal bands will be measured in two-thirds of the total cerebral spinal fluid samples available (n= 121) from patients in the SFSEP, OFSEP and ARISE cohorts by isoelectric focusing.
Aim 2a: Oligoclonal bands as a potential biomarker of RIS. | Week 96
  Oligoclonal bands will be measured in two-thirds of the total cerebral spinal fluid samples available (n= 121) from patients in the SFSEP, OFSEP and ARISE cohorts by isoelectric focusing.
Aim 2b: Validation of cerebrospinal fluid neurofilament light chain as a potential biomarker of RIS. | Week 0
  The neurofilament light chain will be measured in the remaining third of the total cerebral spinal fluid samples available (n= 60) from patients in the SFSEP, OFSEP and ARISE cohorts by isoelectric focusing.
Aim 2b: Validation of cerebrospinal fluid neurofilament light chain as a potential biomarker of RIS. | Week 96
  The neurofilament light chain will be measured in the remaining third of the total cerebral spinal fluid samples available (n= 60) from patients in the SFSEP, OFSEP and ARISE cohorts by isoelectric focusing.
Aim 2b: Validation of chitinase-3-like protein 1 as a potential biomarker of RIS. | Week 0
  Chitinase-3-like protein 1 will be measured in the remaining third of the total cerebral spinal fluid samples available (n=60) from patients in the SFSEP, OFSEP and ARISE cohorts by cytokine multiplex assay (ProcartaPlexTM).
Aim 2b: Validation of chitinase-3-like protein 1 as a potential biomarker of RIS. | Week 96
  Chitinase-3-like protein 1 will be measured in the remaining third of the total cerebral spinal fluid samples available (n=60) from patients in the SFSEP, OFSEP and ARISE cohorts by cytokine multiplex assay (ProcartaPlexTM).
Aim 2b: Validation of oligoclonal bands as a potential biomarker of RIS. | Week 0
  Oligoclonal bands will be measured in the remaining third of the total cerebral spinal fluid samples available (n=60) from patients in the SFSEP, OFSEP and ARISE cohorts by isoelectric focusing.
Aim 2b: Validation of oligoclonal bands as a potential biomarker of RIS. | Week 96
  Oligoclonal bands will be measured in the remaining third of the total cerebral spinal fluid samples available (n=60) from patients in the SFSEP, OFSEP and ARISE cohorts by isoelectric focusing.
Aim 3: Improving prediction of clinical disease activity of RIS | Week 0
  Using patients from Aim 2 (n=181), a multivariate Cox regression model including known predictors of clinical disease activity (sex, age, OCBs, infratentorial and spinal cord lesions, Gd+ lesions, and DMT exposure) will be built to discern the added value of sNfL, sGFAP, and our final set of biomarkers from Aim 2 to predict clinical disease. Biomarker thresholds will be defined based on the distribution of the data.
Aim 3: Improving prediction of clinical disease activity of RIS | Week 96
  Using patients from Aim 2 (n=181), a multivariate Cox regression model including known predictors of clinical disease activity (sex, age, OCBs, infratentorial and spinal cord lesions, Gd+ lesions, and DMT exposure) will be built to discern the added value of sNfL, sGFAP, and our final set of biomarkers from Aim 2 to predict clinical disease. Biomarker thresholds will be defined based on the distribution of the data.

OTHER OUTCOMES:
Age of patients who provided serum and cerebrospinal fluid samples | Week 0
  The ages of patients from the 4 cohorts (ARISE, TERIS, OFSEP and SFSEP) will be recorded in years.
Sex of patients who provided serum and cerebrospinal fluid samples | Week 0
  The sex of patients from the 4 cohorts (ARISE, TERIS, OFSEP and SFSEP) will be recorded as Male/Female/Non-binary.
Disease-Modifying Therapy exposure in patients who provided serum and cerebrospinal fluid samples | Week 0
  Any exposure to disease-modifying therapy among patients from the 4 cohorts (ARISE, TERIS, OFSEP and SFSEP) will be recorded in terms of nature and duration.

CONTACTS AND LOCATIONS:
Locations (3):
- University of Texas, Southwestern, Dallas, Texas, United States
- France (2):
  - COTE D'AZUR UNIVERSITY, URRIS-UR2CA. Hôpital Pasteur 2, 30, Voie Romaine, Nice, Alpes-Maritimes
  - INTERNATIONAL CENTER OF RESEARCH IN INFECTIOLOGY, LYON UNIVERSITY, INSERM U1111, CNRS UMR 5308, ENS, UCBL 46 Allée d'Italie, Lyon, Rhône